CLINICAL TRIAL: NCT04815798
Title: A Randomized, Double-blind Study to Evaluate the Safety, Tolerability, and Potential Efficacy of BACTELIDE vs. Placebo in Addition to Standard-of-care Therapy for S. Aureus, P. Aeruginosa, and K. Pneumoniae Colonized Pressure Injuries
Brief Title: Phage Therapy for the Prevention and Treatment of Pressure Ulcers.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Precisio Biotix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGX-20001
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Pressure Ulcer
Keywords: Wound infection; Pressure injury; Bedsores; Pseudomonas aeruginosa; Klebsiella pneumoniae; Staphylococcus aureus; Resistant infection; Phage; Bacteriophage
MeSH Terms: conditions — Pressure Ulcer; Wound Infection; Pseudomonas Infections; Staphylococcal Infections | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bacteriophage-loaded Microcapsule Spray with Standard of Care (Experimental): Phage therapy (Bacteriophage-loaded Microcapsule Spray) will be administered topically in conjunction with standard of care for pressure ulcers.
  Interventions: Combination Product: Bacteriophage-loaded Microcapsule Spray; Procedure: Standard of Care
- Placebo with Standard of Care (Placebo Comparator): Placebo, analogous to the experimental arm, will be administered topically in conjunction with standard of care for pressure ulcers.
  Interventions: Combination Product: Placebo; Procedure: Standard of Care

INTERVENTIONS:
Combination Product: Bacteriophage-loaded Microcapsule Spray — Study intervention consists of a dosage-metered airless spray containing a cocktail of 14 bacteriophages encapsulated in a biodegradable polymer. This bacteriophage product will be delivered topically every 3 days for 56 days or until wound has healed.
  Other Names: BACTELIDE; PL-03-BM
  Arms: Bacteriophage-loaded Microcapsule Spray with Standard of Care
Combination Product: Placebo — Placebo intervention consists of a dosage-metered airless spray containing a buffer solution analogous to the study intervention. This placebo will be delivered topically every 3 days for 56 days or until wound has healed.
  Arms: Placebo with Standard of Care
Procedure: Standard of Care — Standard of care consists of but is not limited to offloading, positioning, cleansing, debridement, and wound dressing. A topical antimicrobial hydrogel will applied to wounds with signs of localized infection.

SUMMARY:
This study will evaluate a topical bacteriophage therapy product (BACTELIDE) as an adjunct to standard therapy for the prevention and treatment of pressure ulcers colonized with S. aureus, P. aeruginosa, or K. pneumoniae species.

This study will compare the safety and efficacy of BACTELIDE in conjunction with standard of care (SOC) versus a placebo in conjunction with standard of care.

DETAILED DESCRIPTION:
The central aim of this study is to investigate the safety, tolerability, and indicative efficacy of a single dose of a phage therapy combination product, BACTELIDE, as an adjunct to standard therapy in participants presenting with a Stage II, III or IV pressure injuries with positive wound cultures for S. aureus, P. aeruginosa, or K. pneumoniae at screening.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Stated willingness to comply with lifestyle considerations
4. Male or female, 18 years or older presenting in long-term care facilities, out-patient department or in-hospital patients with a stage II, III or IV pressure injury with or without local signs of infection with a size not exceeding 28 cm2
5. Within 72 hours before randomization, pressure injury specimen positive for S. aureus, P. aeruginosa, or K. pneumoniae determined by qPCR or rapid diagnostic test or conventional method or positive growth on specific agar.
6. For females of reproductive potential: use of a highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of administration of the study intervention
7. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.

Exclusion Criteria:

1. Diagnosis of Kennedy terminal ulcer, Trombley-Brennan terminal tissue injuries or skin changes at life's end (SCALE).
2. Pregnancy or lactation.
3. Known allergic reactions to components of SilvaSorb hydrogel.
4. Known allergic reactions to components of the phage treatment; including known allergic reactions to bacteriophages, polyester amide urea polymers and/or TMN buffer.
5. Unstable coronary artery disease.
6. Patients diagnosed with Type I or Type II diabetes, uncontrolled (HgbA1c >8% or 2+ glycosuria).
7. Treatment with another investigational drug or other intervention within 30 days.
8. Intercurrent condition requiring a high dose of chronic corticosteroid therapy, immunosuppressive medication, oncologic chemotherapy.
9. Patients who have additional uncontrolled serious medical or psychiatric illness determined by the investigators where the patient is unfit to receive the product.
10. Chronic stool incontinence without a rectal tube if an individual has a sacral ulcer.
11. Placement of a wound vacuum.
12. Surgical wound closure planned within the study period.
13. Organ failure, acute respiratory failure and chronic renal failure.
14. Diagnosed osteomyelitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events coded by MedDra | At least 56 days
  Safety of BACTELIDE will be measured by the number and percent of treatment related adverse events.
Incidence of treatment discontinuation due to adverse events | 56 days
  Tolerability of BACTELIDE will be measured by the percent premature discontinuation from the study intervention due to treatment emergent Adverse Events

SECONDARY OUTCOMES:
Assess if BACTELIDE can improve the clinical outcome by preventing or treating wound infection. | 28 days
  Response/improvement in treatment-specific clinical outcome based on change in PUSH tool scores.
Assess the effect of BACTELIDE on the incidence of bacterial colonization by S. aureus, P. aeruginosa, or K. pneumoniae species in pressure injury wounds. | 28 days
  Change in the incidence of positive wound cultures for S. aureus, P. aeruginosa, K. pneumoniae collected from surface deep wound swabs and /or tissue specimens.
Assess the effect of BACTELIDE on the rate of wound progression. | 56 days
  Rate of wound progression will be measured by change in viable tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Suh, M.D., Principal Investigator — Mayo Clinic; Karin Zachow, M.D., Principal Investigator — Miami Veterans Affairs Healthcare System; Hector Bolivar, M.D., Principal Investigator — Miami University Health System